CLINICAL TRIAL: NCT04379947
Title: A Real Life All-comers Retrospective Study on FFR-based CABG
Brief Title: Preoperative Use of Fractional Flow Reserve in CABG Use and Effectiveness of FFR-based CABG in Real-life Practice
Status: Withdrawn | Type: Observational
Why Stopped: research group's decision
Sponsor: University of Glasgow (Other)
Responsible Party: Principal Investigator, Cristiano Spadaccio, Clinical Lecturer, University of Glasgow
Other Study IDs: UG-003
Record Dates: First submitted 2020-04-28; First posted 2020-05-08 (Actual); Last update posted 2020-07-13 (Actual); Status verified 2020-07

CONDITIONS: Fracational Flow Reserve; Coronary Artery Disease; Coronary Artery Bypass Surgery
MeSH Terms: conditions — Coronary Artery Disease | interventions — Fractional Flow Reserve, Myocardial

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- FFR-CABG: Patients with at least one intermediate stenosis that received a preoperative FFR evaluation before being referred for CABG
  Interventions: Procedure: Fractional Flow reserve
- Angio-CABG: Patients with at least one intermediate stenosis that did not received a preoperative FFR evaluation before being referred for CABG

INTERVENTIONS:
Procedure: Fractional Flow reserve — Measurement of fractional flow reserve in the preoperative work-up for oronary artery bypass surgery
  Groups: FFR-CABG

SUMMARY:
The use of fractional flow reserve (FFR) to guide coronary artery bypass graft (CABG) is controversial and not ubiquitously adopted across the units. There is no definitive evidence that the use of FFR improves early clinical outcomes after CABG, with the exception of a simplification of the procedure. FFR use may help in defining the indication to the use arterial grafts, but there is no evidence that preoperative FFR lead to any benefits in terms of patency when venous grafts are used.

On these grounds a large multicentric all-comers observational study is planned. The aim is to achieve a real-life picture of the FFR practice in CABG across several European and non-European units. This study will inform on the effective use rate of FFR in the CABG practice and its clinical effectiveness when compared to standard angiography-based CABG.

DETAILED DESCRIPTION:
Background The use of fractional flow reserve (FFR) to guide coronary artery bypass graft (CABG) is controversial. A large retrospective study on 627 patients by Toth et al. showed that FFR-guided surgery was associated with a lower number of graft anastomoses and a lower rate of on-pump surgery compared with angiography-guided coronary artery bypass graft surgery. This did not result in a higher event rate during up to 36 months of follow-up and was associated with a lower rate of angina. The six years follow-up of the same study showed that FFR-guided CABG was associated with a significant reduction in the rate of overall death or myocardial infarction at 6-year follow-up as compared with angiography-guided CABG.

However, the three randomized studies on FFR-based CABG have achieved contradictive results. The FARGO (Fractional Flow Reserve Versus Angiography Randomization for Graft Optimization) and GRAFFITI (GRAft patency after FFR-guided versus angiography-guided CABG) did not report a significant impact on hard outcomes at 1 year. Conversely, the IMPAG trial support the use of preoperative FFR in total arterial CABG. Authors found a significant association between the preoperative FFR measurement of the target vessel and the anastomotic functionality at 6 months, with a cut-off of 0.78. Authors concluded that integration of FFR measurement into the preoperative diagnostic workup could lead to improved anastomotic graft function.

The currently available randomized evidences might have been flawed by limitations including underpowering, entry selectivity bias, cross over among treatment, difference in the type of conduits used and presence of unexpected confounders related to surgeons' reluctance to base their surgical strategy on FFR. These drawbacks not only hamper the reliability of the results, but more importantly, reduce their translatability to the real-life clinical world.

Given the lack of definitive evidences and the difficulty of RCT to capture the real-life scenario of the clinical practice, we plan to perform a large multicentric all-comers study comparing the practice of FFR in CABG across several European and non-European units.

The main aim is to obtain information on

* Use rate of FFR in preoperative planning of surgical candidates
* Effective adherence to FFR guidance during elective surgery and identification of factors eventually limiting observance to FFR information
* Short and long-term outcomes of FFR-based CABG in comparison to standard angiography-based CABG
* Post hoc analysis in relation to type of conduit used, completeness of revascularization, surgeon experience, volume/outcome relationship.

ELIGIBILITY:
Inclusion Criteria:

* all-comers" including both elective and urgent (and urgent in-house) isolated CABG cases

Exclusion Criteria:

* patients undergoing emergency revascularization for iatrogenic complications or other conditions that would prevent a careful analysis of angiographic severity of the lesions

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients will be retrospectively included in the study from 1st December 2010 to 31st December 2019. All surgical candidates with at least one intermediate lesion will be included. Patients that received a preoperative FFR evaluation before being referred for CABG will be part of the FFR-CABG group. The rest of the patients will be included in the Angio-CABG group.
  Inclusion will be on an "all-comers" basis including both elective and urgent (and urgent in-house) isolated CABG cases. However, patients undergoing emergency revascularization for iatrogenic complications or other conditions that would prevent a careful analysis of angiographic severity of the lesions will be excluded.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2020-05 (Estimated); Primary Completion 2020-11 (Estimated); Study Completion 2021-01 (Estimated)

PRIMARY OUTCOMES:
Use rate of FFR in preoperative planning of surgical candidates | 10 years
  Frequency and rate of usage of fractional flow reserve measurement in the routine practice of Cath labs
Effective adherence to FFR guidance during elective surgery and identification of factors eventually limiting observance to FFR information | 10 years
  To check if CABG operations are performed according to the guidance provided by FFR in terms of location and number of lesions to be bypassed
Survival of FFR-based CABG in comparison to standard angiography-based CABG | 10 years
  Comparing mortality rate among the two groups
Myocardial infarction rate in FFR-based CABG in comparison to standard angiography-based CABG | 10 years
  Comparing onset of myocardial infarction among the two groups
Major cardiovascular events rate in FFR-based CABG in comparison to standard angiography-based CABG | 10 years
  Comparing occurrence of major cardiovascular events among the two groups
Target vessel revascularization rate in FFR-based CABG in comparison to standard | 10 years
  Comparing perioperative mortality, myocardial infarction, major cardiovascular events, target vessel revascularization, long-term survival, long-term freedom from coronary intervention among the two groups
Freedom from coronary intervention in FFR-based CABG compared to standard angiography-based CABG | 10 years
  Comparing long-term freedom from coronary intervention among the two groups

SECONDARY OUTCOMES:
Type of conduit used | 10 years
  Post-hoc analysis to investigated the use rate of arterial or venous conduit and the impact on clinical outcomes of the different conduits. This is crucial considering that the most recent randomized trial found a benefit of preoperative FFR when arterial conduits are used for CABG
Completeness of revascularization | 10 years
  to investigate if the use of preoperative FFR is associated to incomplete revascularization (i.e. reduced number of bypassed lesion)
Surgeon experience effect | 10 years
  Measuring relation between surgeon's experience (measured as number of CABG cases performed) on mortality and other outcomes. Studies have demonstrated a learning curve of at least 50 cases
Volume/outcome relationship | 10 years
  Measuring relation between center's experience (measured as number of CABG cases/year) and outcomes.Centers performing high volumes of these procedure might produce better outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Cristiano Spadaccio, MD, PhD, Principal Investigator — University of Glasgow

IPD SHARING:
Plan to Share IPD: No
An anonymous standard data form has been created to retrieve relevant information. The database format along with instruction to insert data in a web-based password-protected database will be provided.

REFERENCES:
- [Background] Sundermann S, Dademasch A, Praetorius J, Kempfert J, Dewey T, Falk V, Mohr FW, Walther T. Comprehensive assessment of frailty for elderly high-risk patients undergoing cardiac surgery. Eur J Cardiothorac Surg. 2011 Jan;39(1):33-7. doi: 10.1016/j.ejcts.2010.04.013. PMID 20627611
- [Background] Coulson TG, Mullany DV, Reid CM, Bailey M, Pilcher D. Measuring the quality of perioperative care in cardiac surgery. Eur Heart J Qual Care Clin Outcomes. 2017 Jan 1;3(1):11-19. doi: 10.1093/ehjqcco/qcw027. PMID 28927188
- [Background] Authors/Task Force members; Windecker S, Kolh P, Alfonso F, Collet JP, Cremer J, Falk V, Filippatos G, Hamm C, Head SJ, Juni P, Kappetein AP, Kastrati A, Knuuti J, Landmesser U, Laufer G, Neumann FJ, Richter DJ, Schauerte P, Sousa Uva M, Stefanini GG, Taggart DP, Torracca L, Valgimigli M, Wijns W, Witkowski A. 2014 ESC/EACTS Guidelines on myocardial revascularization: The Task Force on Myocardial Revascularization of the European Society of Cardiology (ESC) and the European Association for Cardio-Thoracic Surgery (EACTS)Developed with the special contribution of the European Association of Percutaneous Cardiovascular Interventions (EAPCI). Eur Heart J. 2014 Oct 1;35(37):2541-619. doi: 10.1093/eurheartj/ehu278. Epub 2014 Aug 29. No abstract available. PMID 25173339
- [Result] Toth G, De Bruyne B, Casselman F, De Vroey F, Pyxaras S, Di Serafino L, Van Praet F, Van Mieghem C, Stockman B, Wijns W, Degrieck I, Barbato E. Fractional flow reserve-guided versus angiography-guided coronary artery bypass graft surgery. Circulation. 2013 Sep 24;128(13):1405-11. doi: 10.1161/CIRCULATIONAHA.113.002740. Epub 2013 Aug 28. PMID 23985788
- [Result] Fournier S, Toth GG, De Bruyne B, Johnson NP, Ciccarelli G, Xaplanteris P, Milkas A, Strisciuglio T, Bartunek J, Vanderheyden M, Wyffels E, Casselman F, Van Praet F, Stockman B, Degrieck I, Barbato E. Six-Year Follow-Up of Fractional Flow Reserve-Guided Versus Angiography-Guided Coronary Artery Bypass Graft Surgery. Circ Cardiovasc Interv. 2018 Jun;11(6):e006368. doi: 10.1161/CIRCINTERVENTIONS.117.006368. PMID 29848611
- [Result] Thuesen AL, Riber LP, Veien KT, Christiansen EH, Jensen SE, Modrau I, Andreasen JJ, Junker A, Mortensen PE, Jensen LO. Fractional Flow Reserve Versus Angiographically-Guided Coronary Artery Bypass Grafting. J Am Coll Cardiol. 2018 Dec 4;72(22):2732-2743. doi: 10.1016/j.jacc.2018.09.043. PMID 30497559
- [Result] Toth GG, De Bruyne B, Kala P, Ribichini FL, Casselman F, Ramos R, Piroth Z, Fournier S, Piccoli A, Van Mieghem C, Penicka M, Mates M, Nemec P, Van Praet F, Stockman B, Degriek I, Barbato E. Graft patency after FFR-guided versus angiography-guided coronary artery bypass grafting: the GRAFFITI trial. EuroIntervention. 2019 Dec 6;15(11):e999-e1005. doi: 10.4244/EIJ-D-19-00463. PMID 31270037
- [Result] Glineur D, Grau JB, Etienne PY, Benedetto U, Fortier JH, Papadatos S, Laruelle C, Pieters D, El Khoury E, Blouard P, Timmermans P, Ruel M, Chong AY, So D, Chan V, Rubens F, Gaudino MF. Impact of preoperative fractional flow reserve on arterial bypass graft anastomotic function: the IMPAG trial. Eur Heart J. 2019 Aug 1;40(29):2421-2428. doi: 10.1093/eurheartj/ehz329. PMID 31155673
- [Result] Spadaccio C, Glineur D, Barbato E, Di Franco A, Oldroyd KG, Biondi-Zoccai G, Crea F, Fremes SE, Angiolillo DJ, Gaudino M. Fractional Flow Reserve-Based Coronary Artery Bypass Surgery: Current Evidence and Future Directions. JACC Cardiovasc Interv. 2020 May 11;13(9):1086-1096. doi: 10.1016/j.jcin.2019.12.017. Epub 2020 Mar 25. PMID 32222443